CLINICAL TRIAL: NCT02602964
Title: A Randomized Controlled Trial Comparing Deep Versus Moderate Neuromuscular Block - in Low Pressure Pneumoperitoneum - to Optimize the Surgical Conditions During Laparoscopic Donor Nephrectomy
Brief Title: A Trial Comparing Deep Versus Moderate Neuromuscular Block - in Low Pressure Pneumoperitoneum
Acronym: LEOPARD-3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL50874.091.14
Record Dates: First submitted 2015-05-13; First posted 2015-11-11 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-04

CONDITIONS: Nephrostomy; Complications; Pneumoperitoneum; Observation of Neuromuscular Block
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deep neuromsucular block (Experimental): Deep neuromuscular block and low pressure pneumoperitoneum
  Interventions: Other: Deep neuromsucular block
- Standard neuromuscular block (No Intervention): Standard neuromuscular block and low pressure pneumoperitoneum

INTERVENTIONS:
Other: Deep neuromsucular block — Deep or standard neuromuscular block
  Arms: Deep neuromsucular block

SUMMARY:
Live kidney transplantation is first choice for patients with end-stage kidney disease. Therefore, the safety and well-being of kidneys donors are highly important objectives in live kidney donation. Low pressure pneumoperitoneum can decrease postoperative pain and therefore also concomitant use of opioids.

DETAILED DESCRIPTION:
However low pressure pneumoperitoneum can also decrease peri-operative conditions. In this trial the researchers will investigate whether peri-operative conditions during low pressure pneumoperitoneum can be optimized by the use of deep neuromuscular block.

ELIGIBILITY:
Inclusion Criteria:

* obtained informed consent
* age over 18 years

Exclusion Criteria:

* chronic use of analgesics or psychotropic drugs
* use of non-steroidal anti-inflammatory drugs shorter than 5 days before surgery
* known or suspect allergy to rocuronium or sugammadex
* significant liver or renal dysfunction
* pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Mean surgical rating score | perioperative

SECONDARY OUTCOMES:
Conversion to standard pressure pneumoperitoneum | perioperative
Intra-operative complications | perioperative
Length of pneumoperitoneum | perioperative

CONTACTS AND LOCATIONS:
Overall Officials: Denise Özdemir-van Brunschot, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

REFERENCES:
- [Derived] Reijnders-Boerboom GTJA, van Helden EV, Minnee RC, Albers KI, Bruintjes MHD, Dahan A, Martini CH, d'Ancona FCH, Scheffer GJ, Keijzer C, Warle MC. Deep neuromuscular block reduces the incidence of intra-operative complications during laparoscopic donor nephrectomy: a pooled analysis of randomized controlled trials. Perioper Med (Lond). 2021 Dec 9;10(1):56. doi: 10.1186/s13741-021-00224-1. PMID 34879862
- [Derived] Ozdemir-van Brunschot DMD, Braat AE, van der Jagt MFP, Scheffer GJ, Martini CH, Langenhuijsen JF, Dam RE, Huurman VA, Lam D, d'Ancona FC, Dahan A, Warle MC. Deep neuromuscular blockade improves surgical conditions during low-pressure pneumoperitoneum laparoscopic donor nephrectomy. Surg Endosc. 2018 Jan;32(1):245-251. doi: 10.1007/s00464-017-5670-2. Epub 2017 Jun 22. PMID 28643056